CLINICAL TRIAL: NCT00557856
Title: A Phase 1 Pharmacokinetic And Pharmacodynamic Study Of Pf-03446962 In Patients With Advanced Solid Tumors
Brief Title: A First In Patient, Study Of Investigational Drug PF-03446962 In Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A8471001; 2007-001422-27 (EudraCT Number)
Record Dates: First submitted 2007-11-12; First posted 2007-11-14 (Estimated); Results first posted 2015-08-13 (Estimated); Last update posted 2015-10-19 (Estimated); Status verified 2015-09

CONDITIONS: Advanced Solid Tumors
Keywords: Solid Tumors Transforming Growth Factor Beta Activin Receptor-like Kinase 1
MeSH Terms: interventions — ascrinvacumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: PF-03446962

INTERVENTIONS:
Drug: PF-03446962 — To determine the maximum tolerated dose (MTD), and recommended Phase 2 dose (RP2D) of PF-03446962 administered in patients with advanced solid tumors.

SUMMARY:
The purpose of this study is to test the safety and effectiveness of PF-03446962 when given as a single agent. Tumors require new blood vessels to support their ability to grow and to spread (metastasize). New treatments aimed at preventing these blood vessels have the ability to improve the clinical management of cancer.

ELIGIBILITY:
Inclusion Criteria:

* Advanced measurable or non-measurable solid tumors
* Adequate bone marrow function
* Adequate liver function
* Adequate renal function
* Be able and willing to comply with the study scheduled visits, treatment plans, laboratory tests and other procedures

Exclusion Criteria:

* Chemotherapy, radiotherapy, or any investigational cancer therapy within 4 weeks of first dose of study medication
* Active bleeding disorder, including gastrointestinal bleeding, as evidenced by hematemesis, hemoptysis or melena in the past 6 months
* Any of the following within the 12 months prior to starting study treatment: myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass graft, congestive heart failure, cerebrovascular accident including transient ischemic attack, or pulmonary embolus; or any other active thromboembolic event
* QTc prolongation defined as QTc >450 msec
* Patients with known brain metastasis
* Patients with peritoneal carcinosis at risk of bleeding
* Major surgical procedure within 4 weeks of treatment
* Pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2007-11; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (10):
- United States (4):
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Hollings Cancer Center, Charleston, South Carolina
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
- Italy (5):
  - S.C Diagnostica Radiologica 2, Milan
  - S.C. Chirurgia Generale Indirizzo Oncologico 1 (epato-gastro-pancreatica), Milan
  - S.C. Medicina Oncologica I, Fondazione IRCCS Istituto Nazionale Tumori, Milan
  - Dipartimento di Medicina, Milan
  - UO di Oncologia ed Ematologia, Istituto Clinico Humanitas-Humanitas Cancer Center, Rozzano (MI)
- Seoul National University Hospital / Department of Internal Medicine, Seoul, South Korea

REFERENCES:
- [Derived] Simonelli M, Zucali P, Santoro A, Thomas MB, de Braud FG, Borghaei H, Berlin J, Denlinger CS, Noberasco C, Rimassa L, Kim TY, English PA, Abbattista A, Gallo Stampino C, Carpentieri M, Williams JA. Phase I study of PF-03446962, a fully human monoclonal antibody against activin receptor-like kinase-1, in patients with hepatocellular carcinoma. Ann Oncol. 2016 Sep;27(9):1782-7. doi: 10.1093/annonc/mdw240. Epub 2016 Jun 20. PMID 27329247
- [Derived] Goff LW, Cohen RB, Berlin JD, de Braud FG, Lyshchik A, Noberasco C, Bertolini F, Carpentieri M, Stampino CG, Abbattista A, Wang E, Borghaei H. A Phase I Study of the Anti-Activin Receptor-Like Kinase 1 (ALK-1) Monoclonal Antibody PF-03446962 in Patients with Advanced Solid Tumors. Clin Cancer Res. 2016 May 1;22(9):2146-54. doi: 10.1158/1078-0432.CCR-15-1622. Epub 2015 Dec 11. PMID 26655846
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A8471001&StudyName=A%20First%20In%20Patient%2C%20Study%20Of%20Investigational%20Drug%20PF-03446962%20In%20Patients%20With%20Advanced%20Solid%20Tumors

RESULTS

PARTICIPANT FLOW:
Groups:
- PF-03446962 0.5 mg/kg: Part 1: PF-03446962 0.5 milligram per kilogram (mg/kg) intravenous infusion over 1 hour (hr) on Day 1 of cycle 1 (28 days) and on Day 1 of subsequent cycles (14 days) until disease progression, withdrawal by participant or unacceptable toxicity.
- PF-03446962 1 mg/kg: Part 1: PF-03446962 1 mg/kg intravenous infusion over 1 hr on Day 1 of cycle 1 (28 days) and on Day 1 of subsequent cycles (14 days) until disease progression, withdrawal by participant or unacceptable toxicity.
- PF-03446962 2 mg/kg : Part 1: PF-03446962 2 mg/kg intravenous infusion over 1 hr on Day 1 of cycle 1 (28 days) and on Day 1 of subsequent cycles (14 days) until disease progression, withdrawal by participant or unacceptable toxicity.
- PF-03446962 3 mg/kg: Part 1: PF-03446962 3 mg/kg intravenous infusion over 1 hr on Day 1 of cycle 1 (28 days) and on Day 1 of subsequent cycles (14 days) until disease progression, withdrawal by participant or unacceptable toxicity.
- PF-03446962 4.5 mg/kg: Part 1: PF-03446962 4.5 mg/kg intravenous infusion over 1 hr on Day 1 of cycle 1 (28 days) and on Day 1 of subsequent cycles (14 days) until disease progression, withdrawal by participant or unacceptable toxicity.
- PF-03446962 6.75 mg/kg: Part 1: PF-03446962 6.75 mg/kg intravenous infusion over 1 hr on Day 1 of cycle 1 (28 days) and on Day 1 of subsequent cycles (14 days) until disease progression, withdrawal by participant or unacceptable toxicity.
- PF-03446962 10 mg/kg: Part 1: PF-03446962 10 mg/kg intravenous infusion over 1 hr on Day 1 of cycle 1 (28 days) and on Day 1 of subsequent cycles (14 days) until disease progression, withdrawal by participant or unacceptable toxicity.
- PF-03446962 15 mg/kg: Part 1: PF-03446962 15 mg/kg intravenous infusion over 1 hr on Day 1 of cycle 1 (28 days) and on Day 1 of subsequent cycles (14 days) until disease progression, withdrawal by participant or unacceptable toxicity.
- PF-03446962 7 mg/kg: Part 2: PF-03446962 7 mg/kg intravenous infusion over 1 hr on Day 1 of cycle 1 (28 days) and on Day 1 of subsequent cycles (14 days) until disease progression, withdrawal by participant or unacceptable toxicity.
Period: Part 1: Dose Escalation Phase
Arm/Group | PF-03446962 0.5 mg/kg: Part 1 | PF-03446962 1 mg/kg: Part 1 | PF-03446962 2 mg/kg : Part 1 | PF-03446962 3 mg/kg: Part 1 | PF-03446962 4.5 mg/kg: Part 1 | PF-03446962 6.75 mg/kg: Part 1 | PF-03446962 10 mg/kg: Part 1 | PF-03446962 15 mg/kg: Part 1 | PF-03446962 7 mg/kg: Part 2
Started | 7 | 5 | 6 | 3 | 4 | 8 | 7 | 6 | 0
Treated | 5 | 5 | 6 | 3 | 4 | 8 | 7 | 6 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 7 | 5 | 6 | 3 | 4 | 8 | 7 | 6 | 0
Not completed — objective progression or relapse | 3 | 5 | 3 | 1 | 3 | 2 | 5 | 3 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 1 | 1 | 1 | 3 | 1 | 2 | 0
Not completed — Other | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — global deterioration of health status | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0
Not completed — randomized but not treated | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 2: Exploratory Phase
Arm/Group | PF-03446962 0.5 mg/kg: Part 1 | PF-03446962 1 mg/kg: Part 1 | PF-03446962 2 mg/kg : Part 1 | PF-03446962 3 mg/kg: Part 1 | PF-03446962 4.5 mg/kg: Part 1 | PF-03446962 6.75 mg/kg: Part 1 | PF-03446962 10 mg/kg: Part 1 | PF-03446962 15 mg/kg: Part 1 | PF-03446962 7 mg/kg: Part 2
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 24
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 24
Not completed — objective progression or relapse | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 15
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Not completed — global deterioration of health status | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety population included all enrolled participants who received at least one dose of study drug.
Groups:
- PF-03446962: All participants who received PF-03446962 intravenous infusion (0.5 milligram/kilogram [mg/kg], 1 mg/kg, 2 mg, 3 mg/kg, 4.5 mg/kg, 6.75 mg/kg, 10 mg/kg, 15 mg/kg, 7 mg/kg), on Day 1 of cycle 1 (28 days) and on Day 1 of subsequent cycles (14 days) until disease progression or unacceptable toxicity.
Arm/Group | PF-03446962
Number analyzed (Participants) | 68
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.3 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 44

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD): Part 1
Description: MTD was defined as highest dose level for which no more than 1 participant in a dose cohort experienced DLT and at least 2 out of 3/6 participants in the next higher dose. DLT was defined as any of the following events occurring during the first 42 days of study drug: any grade greater than or equal to 3 hematologic and non-hematologic toxicity, all non-disease-related adverse events (AEs).
Time Frame: Baseline up to 42 days after the start of each increased treatment dose
Population: The MTD analysis set included all participants who were enrolled in the dose escalation part of the study and received at least 1 dose of study drug.
Measure: Number; unit: milligram/kilogram (mg/kg)
Groups:
- PF-03446962: All participants who received PF-03446962 intravenous infusion (0.5 milligram/kilogram [mg/kg], 1 mg/kg, 2 mg, 3 mg/kg, 4.5 mg/kg, 6.75 mg/kg, 10 mg/kg, 15 mg/kg), on Day 1 of cycle 1 (28 days) and on Day 1 of subsequent cycles (14 days) until disease progression or unacceptable toxicity.
Arm/Group | PF-03446962
Number analyzed (Participants) | 44
milligram/kilogram (mg/kg) | 10.0

2. Primary Outcome: Recommended Phase 2 Dose (RP2D): Part 1
Description: RP2D was defined as the lower dose level to MTD based on the safety profile.
Time Frame: Baseline up to 42 days after the start of each increased treatment dose
Population: as for outcome 1
Measure: Number; unit: mg/kg
Arm/Group | PF-03446962
Number analyzed (Participants) | 44
mg/kg | 7.0

3. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs): Part 1 and Part 2
Description: An all causality AE was any untoward medical occurrence in participant who received study drug without regard to possibility of causal relationship. Treatment-related AEs was any untoward medical occurrence in participant that was attributed to study drug. Treatment-emergent events were events between first dose of study drug and up to 28 days after last dose that were absent before treatment or that worsened relative to pretreatment state.
Time Frame: Cycle 1 of Day 1 up to 28 days after the last dose of treatment
Population: Safety population included all enrolled participants who received at least one dose of study drug.
Measure: Number; unit: participants
Groups:
- PF-03446962 1 mg/kg: PF-03446962 1 mg/kg intravenous infusion over 1 hr on Day 1 of cycle 1 (28 days) and on Day 1 of subsequent cycles (14 days) until disease progression, withdrawal by participant or unacceptable toxicity.
Arm/Group | PF-03446962 0.5 mg/kg: Part 1 | PF-03446962 1 mg/kg | PF-03446962 2 mg/kg : Part 1 | PF-03446962 3 mg/kg: Part 1 | PF-03446962 4.5 mg/kg: Part 1 | PF-03446962 6.75 mg/kg: Part 1 | PF-03446962 10 mg/kg: Part 1 | PF-03446962 15 mg/kg: Part 1 | PF-03446962 7 mg/kg: Part 2
Number analyzed (Participants) | 5 | 5 | 6 | 3 | 4 | 8 | 7 | 6 | 24
participants
  All causalities | 5 | 5 | 6 | 3 | 4 | 8 | 7 | 6 | 24
  Treatment-related | 4 | 2 | 4 | 1 | 3 | 7 | 6 | 2 | 20

4. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (AEs) Based on Severity: Part 1 and Part 2
Description: AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. AE was assessed according to severity; Grade 0 (no change from normal); grade 1 (mild AE which did not cause any significant problem, no dose adjustment required); grade 2 (moderate AE which caused problem that did not interfere significantly with usual activities or the clinical status, dose adjustment needed due to adverse event); grade 3 (severe AE which caused problem that interfered significantly with usual activities or the clinical status, study drug stopped due to adverse event); grade 4 (life threatening AE) and grade 5 (death). Treatment-emergent events were events between first dose of study drug and up to 28 days after last dose that were absent before treatment or that worsened relative to pretreatment state.
Time Frame: Cycle 1 of Day 1 up to 28 days after the last dose of treatment
Population: Safety population included all enrolled participants who received at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | PF-03446962 0.5 mg/kg: Part 1 | PF-03446962 1 mg/kg: Part 1 | PF-03446962 2 mg/kg : Part 1 | PF-03446962 3 mg/kg: Part 1 | PF-03446962 4.5 mg/kg: Part 1 | PF-03446962 6.75 mg/kg: Part 1 | PF-03446962 10 mg/kg: Part 1 | PF-03446962 15 mg/kg: Part 1 | PF-03446962 7 mg/kg: Part 2
Number analyzed (Participants) | 5 | 5 | 6 | 3 | 4 | 8 | 7 | 6 | 24
participants
  Grade 1 | 3 | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 3
  Grade 2 | 1 | 3 | 1 | 1 | 4 | 3 | 3 | 1 | 7
  Grade 3 | 0 | 0 | 4 | 1 | 0 | 2 | 3 | 3 | 9
  Grade 4 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 4
  Grade 5 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 1

5. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (AEs) Based on Seriousness: Part 1 and Part 2
Description: AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Seriousness of an AE was assessed as serious adverse event (SAE) and non-serious adverse event (non-SAE). An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Non-SAE included all AE minus SAE. Treatment-emergent events were events between first dose of study drug and up to 28 days after last dose that were absent before treatment or that worsened relative to pretreatment state.
Time Frame: Cycle 1 of Day 1 up to 28 days after the last dose of treatment
Population: Safety population included all enrolled participants who received at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | PF-03446962 0.5 mg/kg: Part 1 | PF-03446962 1 mg/kg: Part 1 | PF-03446962 2 mg/kg : Part 1 | PF-03446962 3 mg/kg: Part 1 | PF-03446962 4.5 mg/kg: Part 1 | PF-03446962 6.75 mg/kg: Part 1 | PF-03446962 10 mg/kg: Part 1 | PF-03446962 15 mg/kg: Part 1 | PF-03446962 7 mg/kg: Part 2
Number analyzed (Participants) | 5 | 5 | 6 | 3 | 4 | 8 | 7 | 6 | 24
participants
  Non-Serious Adverse Events | 5 | 5 | 6 | 3 | 4 | 8 | 7 | 6 | 24
  Serious Adverse Events | 2 | 0 | 3 | 0 | 1 | 4 | 2 | 3 | 9

6. Secondary Outcome: Time to Treatment-Emergent Adverse Events (AEs): Part 1 and Part 2
Description: Total time from onset of adverse event till the event is resolved. Treatment-emergent events were events between first dose of study drug and up to 28 days after last dose that were absent before treatment or that worsened relative to pretreatment state.
Time Frame: Cycle 1 of Day 1 up to 28 days after the last dose of treatment
Population: Data for timing was reported in individual participant listing for every adverse event (AE) and mentioned for description of narrative of Serious AEs but was not statistically summarized for analysis on the entire safety population, as planned.
Arm/Group | PF-03446962 0.5 mg/kg: Part 1 | PF-03446962 1 mg/kg: Part 1 | PF-03446962 2 mg/kg : Part 1 | PF-03446962 3 mg/kg: Part 1 | PF-03446962 4.5 mg/kg: Part 1 | PF-03446962 6.75 mg/kg: Part 1 | PF-03446962 10 mg/kg: Part 1 | PF-03446962 15 mg/kg: Part 1 | PF-03446962 7 mg/kg: Part 2
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

7. Secondary Outcome: Number of Participants With Laboratory Abnormalities: Part 1 and Part 2
Description: Laboratory tests included hematology (hemoglobin, lymphocytes absolute [abs], neutrophils abs, platelets, white blood cells) and chemistry (alanine aminotransferase, alkaline phosphatase, amylase, aspartate aminotransferase, bilirubin, creatinine, hypercalcemia, hyperglycemia, hyperkalemia, hypernatremia, hypoalbuminemia, hypocalcemia, hypokalemia, hyponatremia, hypophosphatemia, lipase). Assays were based on National Cancer Institute [NCI] Common Terminology Criteria for AE (CTCAE) grading scale for AEs (grade 1 [mild AE: did not cause any significant problem, no dose adjustment required]; grade 2 [moderate AE: caused problem that did not interfere significantly with usual activities or the clinical status, dose adjustment needed due to adverse event]; grade 3 [severe AE: caused problem that interfered significantly with usual activities or the clinical status, study drug stopped due to adverse event] and grade 4 [life threatening AE]). Overall data of the 4 grades is reported.
Time Frame: Cycle 1 of Day 1 up to 28 days after the last dose of treatment
Population: Safety population included all enrolled participants who received at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | PF-03446962 0.5 mg/kg: Part 1 | PF-03446962 1 mg/kg: Part 1 | PF-03446962 2 mg/kg : Part 1 | PF-03446962 3 mg/kg: Part 1 | PF-03446962 4.5 mg/kg: Part 1 | PF-03446962 6.75 mg/kg: Part 1 | PF-03446962 10 mg/kg: Part 1 | PF-03446962 15 mg/kg: Part 1 | PF-03446962 7 mg/kg: Part 2
Number analyzed (Participants) | 5 | 5 | 6 | 3 | 4 | 7 | 7 | 6 | 24
participants
  Hemoglobin | 4 | 4 | 5 | 1 | 3 | 5 | 4 | 2 | 20
  Lymphocytes abs | 4 | 4 | 4 | 1 | 2 | 4 | 2 | 2 | 12
  Neutrophils abs | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
  Platelets | 1 | 1 | 2 | 2 | 1 | 2 | 3 | 2 | 12
  White blood cells | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 4
  Alanine Aminotransferase | 1 | 0 | 0 | 1 | 1 | 3 | 2 | 5 | 18
  Alkaline Phosphatase | 1 | 3 | 4 | 0 | 3 | 4 | 6 | 6 | 20
  Amylase | 0 | 1 | 3 | 1 | 2 | 2 | 2 | 1 | 6
  Aspartate Aminotransferase | 0 | 0 | 1 | 1 | 2 | 2 | 5 | 5 | 20
  Bilirubin | 0 | 0 | 2 | 1 | 0 | 2 | 2 | 2 | 11
  Creatinine | 1 | 2 | 0 | 2 | 1 | 2 | 3 | 5 | 10
  Hypercalcemia | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 1
  Hyperglycemia | 4 | 3 | 6 | 1 | 4 | 5 | 5 | 4 | 23
  Hyperkalemia | 0 | 0 | 1 | 1 | 0 | 1 | 3 | 0 | 5
  Hypernatremia | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Hypoalbuminemia | 1 | 0 | 2 | 0 | 2 | 4 | 3 | 2 | 12
  Hypocalcemia | 1 | 0 | 1 | 0 | 0 | 1 | 3 | 2 | 6
  Hypokalemia | 2 | 0 | 1 | 0 | 2 | 3 | 0 | 0 | 7
  Hyponatremia | 1 | 1 | 2 | 2 | 2 | 5 | 6 | 5 | 17
  Hypophosphatemia | 1 | 1 | 2 | 1 | 0 | 1 | 2 | 0 | 10
  Lipase | 1 | 1 | 2 | 1 | 1 | 0 | 1 | 2 | 7
  Hypoglycemia | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0

8. Secondary Outcome: Percentage of Participants With Objective Response: Part 1 and Part 2
Description: Percentage of participants with objective response based assessment of confirmed complete response (CR) or confirmed partial response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST). Confirmed responses are those that persist on repeat imaging study at least 4 weeks after initial documentation of response. CR defined as disappearance of all target lesions and non-target lesions. PR defined as >=30 % decrease in sum of the longest diameters (LD) of the target lesions taking as a reference the baseline sum LD according to RECIST associated to non-progressive disease response for non-target lesions.
Time Frame: Baseline then 6 weeks after Cycle 1 of Day1 thereafter every 6 weeks up to Day 490
Population: Response-evaluable set included all participants who received at least 1 dose of study drug with an adequate baseline tumor assessment.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | PF-03446962 0.5 mg/kg: Part 1 | PF-03446962 1 mg/kg: Part 1 | PF-03446962 2 mg/kg : Part 1 | PF-03446962 3 mg/kg: Part 1 | PF-03446962 4.5 mg/kg: Part 1 | PF-03446962 6.75 mg/kg: Part 1 | PF-03446962 10 mg/kg: Part 1 | PF-03446962 15 mg/kg: Part 1 | PF-03446962 7 mg/kg: Part 2
Number analyzed (Participants) | 5 | 5 | 6 | 3 | 4 | 8 | 7 | 6 | 24
percentage of participants | 0 [0.0 to 45.1] | 0 [0.0 to 45.1] | 16.7 [0.9 to 58.2] | 0 [0.0 to 63.2] | 0 [0.0 to 52.7] | 0 [0.0 to 31.2] | 28.6 [5.3 to 65.9] | 0 [0.0 to 39.3] | 0 [0.0 to 11.7]

9. Secondary Outcome: Percentage of Participants With Disease Control: Part 2
Description: Participants who achieved either a confirmed complete Response or confirmed partial response or a Stable disease lasting at least 12 weeks from the first dose was defined as achieving disease control. Confirmed responses are those that persist on repeat imaging study at least 4 weeks after initial documentation of response. CR: disappearance of all target lesions and non-target lesions. PR: >=30 % decrease in sum of the longest diameters (LD) of the target lesions taking as a reference the baseline sum LD and stable disease: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD taking as a reference the smallest sum of the LD according to RECIST associated to non-progressive disease response for non-target lesions. Percentage of participants achieving disease control was calculated out of the participants participating in the exploratory phase.
Time Frame: Baseline then 6 weeks after Cycle 1 of Day1 thereafter every 6 weeks up to Day 490
Population: Response-evaluable set included all participants who started Cycle 1 with an adequate baseline tumor assessment.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | PF-03446962 7 mg/kg: Part 2
Number analyzed (Participants) | 24
percentage of participants | 29.2 [14.6 to 47.9]

10. Secondary Outcome: Time To Progression (TTP): Part 2
Description: Time in months from start of treatment to first documentation of objective tumor progression. TTP was calculated as (first event date or last known progression-free date minus the date of treatment plus 1) divided by 30.44. Tumor progression was determined from oncologic assessment data (where data meet the criteria for progressive disease [PD] per RECIST). PD: >=20% increase in the sum of the LD of the target lesions taking as a reference the smallest sum of the LD or the appearance of one or more new lesions and as unequivocal progression of existing non-target lesions, or the appearance of >=1 new lesions. TTP was calculated out of the participants participating in the exploratory phase.
Time Frame: Baseline then 6 weeks after Cycle 1 of Day1 thereafter every 6 weeks up to Day 490
Population: Safety population included all participants who received at least one dose of study drug.
Measure: Median (Full Range); unit: months
Arm/Group | PF-03446962 7 mg/kg: Part 2
Number analyzed (Participants) | 24
months | 3.0 [1.4 to 4.7]

11. Other Pre Specified Outcome: Maximum Observed Serum Concentration (Cmax): Part 1 and Part 2
Time Frame: 0 hr (pre-dose),0.5,1,1.5,2,5,10,24 hr post-dose on Day (D) 1,3,5,8,11,15,22 of Cycle (C) 1, 0 hr,1 hr post-dose on Day 1 of subsequent cycles up to cycle 12, 28 days after last dose for dose (up to 3 months after last dose for >=2 mg/kg arms)
Population: Pharmacokinetic analysis set included all participants who received at least one dose of study drug and who had complete sampling for pharmacokinetic profiles for PF-03446962.
Measure: Geometric Mean (Standard Deviation); unit: nanogram/milliliter (ng/mL)
Arm/Group | PF-03446962 0.5 mg/kg: Part 1 | PF-03446962 1 mg/kg: Part 1 | PF-03446962 2 mg/kg : Part 1 | PF-03446962 3 mg/kg: Part 1 | PF-03446962 4.5 mg/kg: Part 1 | PF-03446962 6.75 mg/kg: Part 1 | PF-03446962 10 mg/kg: Part 1 | PF-03446962 15 mg/kg: Part 1 | PF-03446962 7 mg/kg: Part 2
Number analyzed (Participants) | 5 | 5 | 6 | 3 | 4 | 8 | 7 | 6 | 24
nanogram/milliliter (ng/mL) | 7210 (2004.0) | 18510 (5623.4) | 38090 (20361) | 62530 (25484) | 123700 (49961) | 140600 (49562) | 274500 (102100) | 304000 (131350) | 153100 (60116)

12. Other Pre Specified Outcome: Minimum Observed Serum Trough Concentration (Cmin): Part 1 and Part 2
Time Frame: 0 hr (pre dose), 1 hr post-dose C1D1, 0 hr,1 hr post-dose on Day 1 of subsequent cycles up to C12
Population: Pharmacokinetic analysis set included all participants who received at least one dose of study drug and who had complete sampling for pharmacokinetic profiles for PF-03446962. Here "N" (Number of participants analyzed) signifies those who were evaluable for the measure and "n" signifies those participants who were evaluable at specific time-point.
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | PF-03446962 0.5 mg/kg: Part 1 | PF-03446962 1 mg/kg: Part 1 | PF-03446962 2 mg/kg : Part 1 | PF-03446962 3 mg/kg: Part 1 | PF-03446962 4.5 mg/kg: Part 1 | PF-03446962 6.75 mg/kg: Part 1 | PF-03446962 10 mg/kg: Part 1 | PF-03446962 15 mg/kg: Part 1 | PF-03446962 7 mg/kg: Part 2
Number analyzed (Participants) | 3 | 2 | 6 | 3 | 4 | 5 | 5 | 2 | 15
ng/mL
  Cycle 2 Day 1 (n=3, 2, 6, 3, 4, 5, 5, 2, 15) | NA (NA) — Data was not analyzed since no participants were evaluable for at this time point for the specific arm group. | NA (NA) — Data was not analyzed since no participants were evaluable for at this time point for the specific arm group. | 1010 (1377.1) | 4473 (1888.6) | 8675 (2203.0) | 14820 (4943.4) | 33440 (14738) | 35450 (1060.7) | 17230 (8815.0)
  Cycle 3 Day 1 (n=3, 2, 4, 3, 1, 4, 3, 1, 13) | NA (NA) — Data was not analyzed since no participants were evaluable for at this time point for the specific arm group. | 704.0 (461.03) | 9992 (14932) | 17070 (5122.8) | 4850 (NA) — Standard deviation was not reported since only 1 participant was evaluable for this arm group. | 45850 (15660) | 77530 (31351) | 69400 (NA) — Standard deviation was not reported since only 1 participant was evaluable for this arm group. | 40870 (25784)
  Cycle 4 Day 1 (n=2, 2, 2, 3, 1, 4, 3, 1, 12) | NA (NA) — Data was not analyzed since no participants were evaluable for at this time point for the specific arm group. | 2000 (353.55) | 6715 (2934.5) | 22030 (3931.1) | 32700 (NA) — Standard deviation was not reported since only 1 participant was evaluable for this arm group. | 41880 (3108.5) | 93130 (44384) | 87100 (NA) — Standard deviation was not reported since only 1 participant was evaluable for this arm group. | 64960 (35284)
  Cycle 5 Day 1 (n= 1, 0, 2, 3, 1, 3, 3, 1, 12) | 588.0 (NA) — Standard deviation was not reported since only 1 participant was evaluable for this arm group. | NA (NA) — Data was not analyzed since no participants were evaluable for at this time point for the specific arm group. | 11490 (3691.1) | 25930 (5488.5) | 42200 (NA) — Standard deviation was not reported since only 1 participant was evaluable for this arm group. | 51600 (12065) | 103300 (56589) | 98800 (NA) — Standard deviation was not reported since only 1 participant was evaluable for this arm group. | 76960 (40711)
  Cycle 6 Day 1 (n=0, 2, 2, 1, 1, 1, 1, 0, 7) | NA (NA) — Data was not analyzed since no participants were evaluable for at this time point for the specific arm group. | NA (NA) — Data was not analyzed since no participants were evaluable for at this time point for the specific arm group. | 13470 (6554.9) | NA (NA) — Data was not analyzed since no participants were evaluable for at this time point for the specific arm group. | 45000 (NA) — Standard deviation was not reported since only 1 participant was evaluable for this arm group. | 58070 (8471.9) | 44700 (NA) — Standard deviation was not reported since only 1 participant was evaluable for this arm group. | NA (NA) — Data was not analyzed since no participants were evaluable for at this time point for the specific arm group. | 69250 (52222)
  Cycle 7 Day 1 (n=0, 0, 2, 1, 1, 3, 1, 0, 7) | NA (NA) — Data was not analyzed since no participants were evaluable for at this time point for the specific arm group. | NA (NA) — Data was not analyzed since no participants were evaluable for at this time point for the specific arm group. | 11920 (7749.9) | 34200 (NA) — Standard deviation was not reported since only 1 participant was evaluable for this arm group. | 45000 (NA) — Standard deviation was not reported since only 1 participant was evaluable for this arm group. | 73670 (24393) | 44700 (NA) — Standard deviation was not reported since only 1 participant was evaluable for this arm group. | NA (NA) — Data was not analyzed since no participants were evaluable for at this time point for the specific arm group. | 68100 (56580)
  Cycle 8 Day 1 (n=0, 0, 2, 1, 1, 2, 1, 0, 5) | NA (NA) — Data was not analyzed since no participants were evaluable for at this time point for the specific arm group. | NA (NA) — Data was not analyzed since no participants were evaluable for at this time point for the specific arm group. | 10850 (353.55) | 43400 (NA) — Standard deviation was not reported since only 1 participant was evaluable for this arm group. | 45100 (NA) — Standard deviation was not reported since only 1 participant was evaluable for this arm group. | 76950 (42497) | 217000 (NA) — Standard deviation was not reported since only 1 participant was evaluable for this arm group. | NA (NA) — Data was not analyzed since no participants were evaluable for at this time point for the specific arm group. | 99740 (66263)
  Cycle 9 Day 1 (n=0, 0, 2, 1, 1, 2, 1, 0, 4) | NA (NA) — Data was not analyzed since no participants were evaluable for at this time point for the specific arm group. | NA (NA) — Data was not analyzed since no participants were evaluable for at this time point for the specific arm group. | 14150 (1626.3) | 47500 (NA) — Standard deviation was not reported since only 1 participant was evaluable for this arm group. | 55200 (NA) — Standard deviation was not reported since only 1 participant was evaluable for this arm group. | 55150 (11526) | 294000 (NA) — Standard deviation was not reported since only 1 participant was evaluable for this arm group. | NA (NA) — Data was not analyzed since no participants were evaluable for at this time point for the specific arm group. | 85750 (57225)
  Cycle 10 Day 1 (n=0, 0, 1, 1, 1, 2, 1, 0, 3) | NA (NA) — Data was not analyzed since no participants were evaluable for at this time point for the specific arm group. | NA (NA) — Data was not analyzed since no participants were evaluable for at this time point for the specific arm group. | 20100 (NA) — Standard deviation was not reported since only 1 participant was evaluable for this arm group. | 43200 (NA) — Standard deviation was not reported since only 1 participant was evaluable for this arm group. | 39000 (NA) — Standard deviation was not reported since only 1 participant was evaluable for this arm group. | 59050 (16334) | 190000 (NA) — Standard deviation was not reported since only 1 participant was evaluable for this arm group. | NA (NA) — Data was not analyzed since no participants were evaluable for at this time point for the specific arm group. | 66620 (50809)
  Cycle 11 Day 1 (n=0, 0, 0, 1, 1, 2, 1, 0, 3) | NA (NA) — Data was not analyzed since no participants were evaluable for at this time point for the specific arm group. | NA (NA) — Data was not analyzed since no participants were evaluable for at this time point for the specific arm group. | NA (NA) — Data was not analyzed since no participants were evaluable for at this time point for the specific arm group. | 44200 (NA) — Standard deviation was not reported since only 1 participant was evaluable for this arm group. | 40500 (NA) — Standard deviation was not reported since only 1 participant was evaluable for this arm group. | 55050 (10677) | 186000 (NA) — Data was not analyzed since no participants were evaluable for at this time point for the specific arm group. | NA (NA) — Data was not analyzed since no participants were evaluable for at this time point for the specific arm group. | 103600 (78883)
  Cycle 12 Day 1 (n=0, 0, 0, 0, 1, 2, 1, 0, 2) | NA (NA) — Data was not analyzed since no participants were evaluable for at this time point for the specific arm group. | NA (NA) — Data was not analyzed since no participants were evaluable for at this time point for the specific arm group. | NA (NA) — Data was not analyzed since no participants were evaluable for at this time point for the specific arm group. | NA (NA) — Data was not analyzed since no participants were evaluable for at this time point for the specific arm group. | 64500 (NA) — Standard deviation was not reported since only 1 participant was evaluable for this arm group. | 52100 (7636.8) | 222000 (NA) — Standard deviation was not reported since only 1 participant was evaluable for this arm group. | NA (NA) — Data was not analyzed since no participants were evaluable for at this time point for the specific arm group. | 69200 (71842)

13. Other Pre Specified Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) of PF-03446962: Part 1 and Part 2
Time Frame: as for outcome 11
Population: Pharmacokinetic analysis set included all participants who received at least one dose of study drug and who had complete sampling for pharmacokinetic profiles for PF-03446962. Here "N" (Number of participants analyzed) signifies those who were evaluable for the measure.
Measure: Median (Full Range); unit: hour
Arm/Group | PF-03446962 0.5 mg/kg: Part 1 | PF-03446962 1 mg/kg: Part 1 | PF-03446962 2 mg/kg : Part 1 | PF-03446962 3 mg/kg: Part 1 | PF-03446962 4.5 mg/kg: Part 1 | PF-03446962 6.75 mg/kg: Part 1 | PF-03446962 10 mg/kg: Part 1 | PF-03446962 15 mg/kg: Part 1 | PF-03446962 7 mg/kg: Part 2
Number analyzed (Participants) | 5 | 5 | 6 | 3 | 4 | 7 | 7 | 5 | 24
hour | 1.50 [1.00 to 2.00] | 1.58 [1.00 to 2.00] | 1.75 [0.917 to 2.50] | 1.50 [1.00 to 2.00] | 1.99 [1.00 to 3.75] | 1.75 [1.17 to 5.00] | 1.50 [0.517 to 5.00] | 3.34 [1.00 to 24.0] | 1.77 [0.900 to 215]

14. Other Pre Specified Outcome: Area Under the Curve From Time Zero to Day 28 [AUC (0-28)]: Part 1 and Part 2
Description: AUC (0-28) = Area under the plasma concentration versus time curve from time zero (pre-dose) to Day 28 (0-28).
Time Frame: as for outcome 11
Population: as for outcome 13
Measure: Geometric Mean (Standard Deviation); unit: nanogram*hour/milliliter (ng*hr/mL)
Arm/Group | PF-03446962 0.5 mg/kg: Part 1 | PF-03446962 1 mg/kg: Part 1 | PF-03446962 2 mg/kg : Part 1 | PF-03446962 3 mg/kg: Part 1 | PF-03446962 4.5 mg/kg: Part 1 | PF-03446962 6.75 mg/kg: Part 1 | PF-03446962 10 mg/kg: Part 1 | PF-03446962 15 mg/kg: Part 1 | PF-03446962 7 mg/kg: Part 2
Number analyzed (Participants) | 5 | 5 | 6 | 3 | 4 | 7 | 7 | 5 | 24
nanogram*hour/milliliter (ng*hr/mL) | 490000 (132220) | 1752000 (436440) | 3281000 (1817700) | 8247000 (2657400) | 15070000 (1447700) | 22890000 (7372200) | 45750000 (15972000) | 52660000 (29315000) | 22890000 (10395000)

15. Other Pre Specified Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast): Part 1 and Part 2
Description: Area under the plasma concentration time-curve from zero to the last measured concentration (AUClast).
Time Frame: as for outcome 11
Population: as for outcome 13
Measure: Geometric Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | PF-03446962 0.5 mg/kg: Part 1 | PF-03446962 1 mg/kg: Part 1 | PF-03446962 2 mg/kg : Part 1 | PF-03446962 3 mg/kg: Part 1 | PF-03446962 4.5 mg/kg: Part 1 | PF-03446962 6.75 mg/kg: Part 1 | PF-03446962 10 mg/kg: Part 1 | PF-03446962 15 mg/kg: Part 1 | PF-03446962 7 mg/kg: Part 2
Number analyzed (Participants) | 5 | 5 | 6 | 3 | 4 | 7 | 7 | 5 | 24
ng*hr/mL | 471400 (124340) | 1683000 (435490) | 3273000 (1819200) | 8247000 (2657400) | 15690000 (2965800) | 21380000 (7823700) | 44110000 (15577000) | 51160000 (21718000) | 22850000 (10504000)

16. Other Pre Specified Outcome: Systemic Clearance(CL): Part 1 and Part 2
Description: CL is a quantitative measure of the rate at which a drug substance is removed from the body. As per planned analysis, CL was summarized if at least 3 participants had reportable value.
Time Frame: as for outcome 11
Population: as for outcome 13
Measure: Geometric Mean (Standard Deviation); unit: liter/hour (L/hr)
Arm/Group | PF-03446962 0.5 mg/kg: Part 1 | PF-03446962 1 mg/kg: Part 1 | PF-03446962 2 mg/kg : Part 1 | PF-03446962 3 mg/kg: Part 1 | PF-03446962 4.5 mg/kg: Part 1 | PF-03446962 6.75 mg/kg: Part 1 | PF-03446962 10 mg/kg: Part 1 | PF-03446962 15 mg/kg: Part 1 | PF-03446962 7 mg/kg: Part 2
Number analyzed (Participants) | 5 | 4 | 6 | 1 | 2 | 3 | 3 | 3 | 7
liter/hour (L/hr) | 0.07675 (0.02318) | 0.03469 (0.00866) | 0.04198 (0.03927) | NA (NA) — Data was not summarized since only 1 participant had reportable value, as per planned analysis. | NA (NA) — Data was not summarized since only 2 participants had reportable value, as per planned analysis. | 0.01861 (0.00225) | 0.01668 (0.00482) | 0.01169 (0.01288) | 0.01921 (0.00507)

17. Secondary Outcome: Volume of Distribution: Part 1 and Part 2
Description: Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired blood concentration of a drug. As per planned analysis, volume of distribution was summarized if at least 3 participants had reportable value.
Time Frame: as for outcome 11
Population: as for outcome 13
Measure: Geometric Mean (Standard Deviation); unit: liter (L)
Arm/Group | PF-03446962 0.5 mg/kg: Part 1 | PF-03446962 1 mg/kg: Part 1 | PF-03446962 2 mg/kg : Part 1 | PF-03446962 3 mg/kg: Part 1 | PF-03446962 4.5 mg/kg: Part 1 | PF-03446962 6.75 mg/kg: Part 1 | PF-03446962 10 mg/kg: Part 1 | PF-03446962 15 mg/kg: Part 1 | PF-03446962 7 mg/kg: Part 2
Number analyzed (Participants) | 5 | 4 | 6 | 1 | 2 | 3 | 3 | 3 | 7
liter (L) | 6.350 (1.1399) | 5.770 (1.1850) | 7.421 (2.8525) | NA (NA) — Data was not summarized since only 1 participant had reportable value, as per planned analysis. | NA (NA) — Data was not summarized since only 2 participants had reportable value, as per planned analysis. | 6.718 (1.2400) | 5.373 (0.85541) | 6.675 (2.4858) | 6.110 (1.6303)

18. Other Pre Specified Outcome: Plasma Decay Half-Life (t1/2): Part 1 and Part 2
Description: Plasma decay half-life is the time measured for the plasma concentration to decrease by one half. As per planned analysis, t1/2 was summarized if at least 3 participants had reportable value.
Time Frame: as for outcome 11
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | PF-03446962 0.5 mg/kg: Part 1 | PF-03446962 1 mg/kg: Part 1 | PF-03446962 2 mg/kg : Part 1 | PF-03446962 3 mg/kg: Part 1 | PF-03446962 4.5 mg/kg: Part 1 | PF-03446962 6.75 mg/kg: Part 1 | PF-03446962 10 mg/kg: Part 1 | PF-03446962 15 mg/kg: Part 1 | PF-03446962 7 mg/kg: Part 2
Number analyzed (Participants) | 5 | 4 | 6 | 1 | 2 | 3 | 3 | 3 | 7
hours | 2.678 (1.0622) | 5.588 (2.3790) | 7.360 (4.5596) | NA (NA) — Data was not summarized since only 1 participant had reportable value, as per planned analysis. | NA (NA) — Data was not summarized since only 2 participants had reportable value, as per planned analysis. | 11.90 (0.88882) | 10.22 (2.3394) | 17.77 (5.6589) | 9.616 (2.3870)

19. Other Pre Specified Outcome: Human Anti - Human Antibody (HAHA) Concentration: Part 1 and Part 2
Description: HAHA concentration was analyzed in blood samples for the evaluation of immunogenicity of PF-03446962. HAHA concentration was reported for samples above lower limit of quantification (>=4.32).
Time Frame: Baseline up to 3 months after last dose
Population: Statistical Data was not statistically summarized as majority of participants had concentration below the limit of quantification.
Arm/Group | PF-03446962 0.5 mg/kg: Part 1 | PF-03446962 1 mg/kg: Part 1 | PF-03446962 2 mg/kg : Part 1 | PF-03446962 3 mg/kg: Part 1 | PF-03446962 4.5 mg/kg: Part 1 | PF-03446962 6.75 mg/kg: Part 1 | PF-03446962 10 mg/kg: Part 1 | PF-03446962 15 mg/kg: Part 1 | PF-03446962 7 mg/kg: Part 2
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

20. Other Pre Specified Outcome: Soluble Protein Biomarker [Angiopoietin-2 (Ang-2), Bone Morphogenetic Protein-9 (BMP-9), Chemokine (C-C Motif) Ligand 2 (CCL2)]: Part 1 and Part 2
Description: Plasma concentrations of soluble proteins (Ang-2, BMP-9, C-C motif) may be associated with tumor angiogenesis or tumor physiology and may correlate with efficacy or biological activity.
Time Frame: Baseline (pre-dose of C1D1), C1D1 6 hours post dosing, C1D22, C2D1, C3D1 and end of treatment (Day 490)
Population: Soluble protein biomarker analysis set included all participants who received at least one dose of study drug with a baseline (pre-dose C1D1) or screening biomarker result, and at least one on-treatment biomarker result for at least one biomarker. "n" signifies those participants who were evaluable at specific time-point.
Measure: Mean (Standard Deviation); unit: picogram/milliliter (pg/mL)
Arm/Group | PF-03446962 0.5 mg/kg: Part 1 | PF-03446962 1 mg/kg: Part 1 | PF-03446962 2 mg/kg : Part 1 | PF-03446962 3 mg/kg: Part 1 | PF-03446962 4.5 mg/kg: Part 1 | PF-03446962 6.75 mg/kg: Part 1 | PF-03446962 10 mg/kg: Part 1 | PF-03446962 15 mg/kg: Part 1 | PF-03446962 7 mg/kg: Part 2
Number analyzed (Participants) | 5 | 5 | 6 | 3 | 4 | 8 | 7 | 6 | 24
picogram/milliliter (pg/mL)
  Baseline: Ang-2 (n=5, 5, 6, 3, 4, 8, 7, 6, 24) | 280.9 (107.01) | 245.2 (85.36) | 405.3 (171.82) | 233.8 (47.89) | 554.3 (404.80) | 629.7 (265.33) | 566.3 (617.76) | 600.5 (469.09) | 1497.4 (881.71)
  C1D16H: Ang-2 (n=4, 3, 6, 3, 4, 8, 7, 6, 24) | 357.7 (87.87) | 326.0 (122.58) | 410.2 (170.55) | 266.3 (28.31) | 580.3 (485.49) | 558.0 (249.90) | 498.4 (508.76) | 548.1 (324.70) | 1509.6 (813.06)
  C1D22: Ang-2 (n=4, 5, 6, 3, 4, 6, 7, 5, 20) | 297.0 (146.98) | 429.8 (202.03) | 489.7 (235.28) | 248.0 (84.73) | 725.2 (654.99) | 491.8 (236.61) | 613.0 (627.25) | 400.0 (198.85) | 1651.4 (894.33)
  C2D1: Ang-2 (n=3, 2, 6, 3, 4, 5, 5, 2, 20) | 304.4 (126.39) | 312.4 (195.37) | 501.2 (194.40) | 205.7 (48.10) | 637.5 (535.52) | 445.3 (231.91) | 557.9 (575.66) | 338.1 (84.57) | 1473.5 (690.55)
  C3D1: Ang-2 (n=3, 2, 4, 3, 1, 4, 3, 1, 12) | 309.1 (133.43) | 338.1 (235.11) | 417.6 (192.35) | 258.3 (57.44) | 501.3 (NA) — Standard deviation was not reported since only 1 participant was evaluable for this arm group. | 510.0 (305.51) | 254.5 (44.89) | 586.8 (NA) — Standard deviation was not reported since only 1 participant was evaluable for this arm group. | 1539.3 (1036.24)
  EOT: Ang-2 (n=5, 5, 2, 3, 4, 4, 5, 5, 17) | 507.2 (375.16) | 355.6 (166.32) | 439.5 (292.25) | 346.7 (57.94) | 775.6 (618.41) | 499.8 (368.96) | 974.9 (1014.67) | 737.9 (572.30) | 2791.2 (3637.55)
  Baseline: BMP-9 (n=5, 5, 6, 3, 4, 8, 7, 6, 24) | 41.7 (44.60) | 18.3 (6.92) | 67.2 (114.87) | 18.4 (11.54) | 68.2 (79.58) | 262.0 (669.08) | 48.9 (23.13) | 29.0 (11.38) | 47.6 (50.88)
  C1D16H: BMP-9 (n=4, 3, 6, 2, 4, 7, 7, 6, 23) | 55.3 (66.60) | 19.5 (10.38) | 56.4 (104.06) | 20.9 (10.39) | 54.1 (58.18) | 273.3 (658.58) | 35.6 (25.63) | 14.0 (5.99) | 45.0 (48.97)
  C1D22: BMP-9 (n=4, 5, 6, 2, 4, 5, 7, 5, 19) | 45.7 (51.45) | 16.7 (7.57) | 60.5 (121.98) | 17.1 (9.90) | 35.7 (36.66) | 394.0 (852.68) | 33.0 (20.44) | 22.0 (12.27) | 39.2 (40.88)
  C2D1: BMP-9 (n=3, 2, 6, 2, 4, 4, 5, 2, 20) | 47.5 (52.77) | 23.9 (0.49) | 54.7 (112.92) | 18.2 (0.28) | 58.9 (85.35) | 391.7 (755.57) | 26.5 (16.89) | 12.2 (4.88) | 40.0 (51.36)
  C3D1: BMP-9 (n=2, 2, 4, 2, 1, 3, 3, 1, 12) | 80.4 (86.41) | 21.3 (2.76) | 99.4 (176.84) | 18.8 (0.00) | 10.8 (NA) — Standard deviation was not reported since only 1 participant was evaluable for this arm group. | 933.3 (1593.69) | 32.2 (13.14) | 16.6 (NA) — Standard deviation was not reported since only 1 participant was evaluable for this arm group. | 40.8 (36.65)
  EOT: BMP-9 (n=5, 5, 2, 2, 4, 4, 5, 5, 17) | 53.2 (70.27) | 15.5 (5.86) | 156.4 (179.39) | 16.5 (2.33) | 75.5 (94.07) | 246.1 (460.69) | 44.0 (35.00) | 17.1 (7.69) | 33.8 (27.55)
  Baseline: CCL2 (n=5, 5, 6, 3, 4, 8, 7, 6, 24) | 1048.4 (259.96) | 897.1 (414.25) | 1296.3 (629.37) | 1179.8 (597.43) | 858.5 (697.41) | 1648.5 (744.80) | 1798.7 (1374.40) | 2659.5 (1356.79) | 1743.1 (1267.52)
  C1D16H: CCL2 (n=4, 3, 6, 3, 4, 8, 7, 6, 24) | 1413.1 (451.52) | 868.2 (348.23) | 1019.8 (222.52) | 845.5 (309.44) | 746.4 (330.31) | 910.1 (297.10) | 1176.7 (198.86) | 1253.9 (353.28) | 887.7 (411.38)
  C1D22: CCL2 (n=4, 5, 6, 3, 4, 6, 7, 5, 20) | 1300.7 (519.44) | 882.1 (300.21) | 1065.6 (491.41) | 898.4 (144.11) | 801.0 (432.10) | 896.0 (365.37) | 1146.9 (400.30) | 1061.8 (469.42) | 846.5 (524.84)
  C2D1: CCL2 (n=3, 2, 6, 3, 4, 5, 5, 2, 20) | 1466.4 (510.75) | 1156.6 (493.42) | 1091.0 (317.65) | 777.6 (220.42) | 692.5 (216.16) | 1206.5 (443.00) | 858.6 (165.26) | 1060.8 (577.85) | 801.9 (338.56)
  C3D1: CCL2 (n=3, 2, 4, 3, 1, 4, 3, 1, 12) | 1413.8 (651.34) | 933.3 (259.79) | 951.0 (418.52) | 793.2 (180.32) | 735.7 (NA) — Standard deviation was not reported since only 1 participant was evaluable for this arm group. | 818.3 (422.89) | 909.9 (278.50) | 617.1 (NA) — Standard deviation was not reported since only 1 participant was evaluable for this arm group. | 791.3 (364.58)
  EOT: CCL2 (n=5, 5, 2, 3, 4, 4, 5, 5, 17) | 1132.1 (202.68) | 898.5 (270.19) | 729.7 (242.18) | 645.4 (94.59) | 699.6 (372.50) | 1190.4 (675.67) | 1176.2 (699.03) | 1179.9 (370.44) | 743.7 (314.64)

21. Other Pre Specified Outcome: Soluble Protein Biomarker [Cluster of Differentiation 106 (CD106), Cluster of Differentiation 54 (CD54), Endoglin]: Part 1 and Part 2
Description: Plasma concentrations of soluble proteins (CD106, CD54 and Endoglin) may be associated with tumor angiogenesis or tumor physiology and may correlate with efficacy or biological activity.
Time Frame: Baseline (pre-dose of C1D1), C1D1 6 hours post dosing, C1D22, C2D1, C3D1 and end of treatment (Day 490)
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | PF-03446962 0.5 mg/kg: Part 1 | PF-03446962 1 mg/kg: Part 1 | PF-03446962 2 mg/kg : Part 1 | PF-03446962 3 mg/kg: Part 1 | PF-03446962 4.5 mg/kg: Part 1 | PF-03446962 6.75 mg/kg: Part 1 | PF-03446962 10 mg/kg: Part 1 | PF-03446962 15 mg/kg: Part 1 | PF-03446962 7 mg/kg: Part 2
Number analyzed (Participants) | 5 | 5 | 6 | 3 | 4 | 8 | 7 | 6 | 24
pg/ml
  Baseline: CD106 (n= 5, 5, 6, 3, 4, 8, 7, 6, 24) | 1426995 (59227.1) | 1977059 (278968) | 2103430 (918193) | 1550000 (637320) | 2317802 (1217870) | 2537306 (1097384) | 1994549 (1151754) | 2380621 (1221978) | 4618397 (2077485)
  C1D16H: CD106 (n= 4, 3, 6, 3, 4, 8, 7, 6, 24) | 1553640 (248023) | 1751998 (131286) | 1997949 (699820) | 1409035 (308143) | 2058998 (1253058) | 2121253 (675955) | 1825721 (1290987) | 2105192 (1365510) | 4441245 (2178832)
  C1D22: CD106 (n= 4, 5, 6, 3, 4, 6, 7, 5, 20) | 1531678 (249394) | 2134392 (357871) | 2251447 (517132) | 1370676 (329573) | 2817598 (2026342) | 2762433 (1722911) | 2701837 (1710834) | 2456276 (1404983) | 5453614 (2116043)
  C2D1: CD106 (n= 3, 2, 6, 3, 4, 5, 5, 2, 20) | 1577290 (378509) | 1799035 (695018) | 2229424 (469152) | 1269574 (366430) | 2370883 (1278663) | 2542120 (2147151) | 1676349 (691658) | 3247890 (1683551) | 5217619 (2747474)
  C3D1: CD106 (n= 3, 2, 4, 3, 1, 4, 3, 1, 12) | 1508775 (201658) | 1994588 (266837) | 2465890 (1070226) | 1892928 (571192) | 2162501 (NA) — Standard deviation was not reported since only 1 participant was evaluable for this arm group. | 3009982 (2128505) | 1380137 (234263) | 4814239 (NA) — Standard deviation was not reported since only 1 participant was evaluable for this arm group. | 4482748 (2376204)
  EOT: CD106 (n= 5, 5, 2, 3, 4, 4, 5, 5, 17) | 2097201 (582243) | 1782709 (473363) | 3480129 (1753142) | 1600889 (484412) | 3004218 (2225879) | 2169361 (755936) | 3869570 (2242247) | 2600730 (1098325) | 6321592 (2385497)
  Baseline: CD54 (n= 5, 5, 6, 3, 4, 8, 7, 6, 24) | 456653 (100191) | 592276 (164098) | 598761 (333166) | 703255 (486462) | 590523 (144561) | 567736 (306989) | 627494 (279501) | 554785 (201270) | 925590 (408338)
  C1D16H: CD54 (n= 4, 3, 6, 3, 4, 8, 7, 6, 24) | 458194 (64789.1) | 512402 (81155.7) | 624061 (233499) | 450887 (168300) | 538807 (172168) | 548456 (201218) | 603467 (311056) | 517460 (251249) | 1053926 (491420)
  C1D22: CD54 (n= 4, 5, 6, 3, 4, 6, 7, 5, 20) | 428766 (80302.4) | 585405 (46397.3) | 578775 (246897) | 356495 (54530.0) | 565451 (196841) | 612504 (370207) | 939357 (706017) | 604023 (291355) | 1173444 (546999)
  C2D1: CD54 (n= 3, 2, 6, 3, 4, 5, 5, 2, 20) | 433203 (90282.8) | 841543 (568591) | 585420 (308551) | 375141 (32483.6) | 628011 (242437) | 575469 (392901) | 641992 (351793) | 727099 (302728) | 980791 (354159)
  C3D1: CD54 (n= 3, 2, 4, 3, 1, 4, 3, 1, 12) | 495252 (112929) | 566407 (160088) | 646360 (390594) | 474589 (70371.2) | 605375 (NA) — Standard deviation was not reported since only 1 participant was evaluable for this arm group. | 664537 (533228) | 414291 (147170) | 890980 (NA) — Standard deviation was not reported since only 1 participant was evaluable for this arm group. | 969068 (433245)
  EOT: CD54 (n= 5, 5, 2, 3, 4, 4, 5, 5, 17) | 535193 (116435) | 504828 (53486.9) | 1022507 (841417) | 483216 (158483) | 600281 (94835.6) | 537001 (171132) | 1096693 (941040) | 569412 (121592) | 1108796 (416355)
  Baseline: Endoglin (n= 5, 5, 6, 3, 4, 8, 7, 6, 24) | 24345.9 (1067.46) | 28133.0 (5202.28) | 22355.2 (5984.52) | 30265.3 (2727.69) | 26342.4 (2922.41) | 24864.6 (3830.51) | 26313.7 (6449.03) | 25599.5 (7530.00) | 32680.3 (6820.09)
  C1D16H: Endoglin (n= 4, 3, 6, 3, 4, 8, 7, 6, 24) | 24961.0 (2310.44) | 24983.9 (5489.16) | 21789.5 (3978.18) | 31365.1 (3547.94) | 25209.2 (3357.89) | 24336.6 (3196.96) | 25110.6 (8066.23) | 26774.1 (11443.0) | 33976.7 (9156.44)
  C1D22: Endoglin (n= 4, 5, 6, 3, 4, 6, 7, 5, 20) | 25412.5 (2910.37) | 30123.0 (2225.81) | 27615.3 (9426.55) | 32203.6 (5574.70) | 26231.6 (3899.05) | 29895.0 (2248.59) | 33397.7 (13366.3) | 24970.6 (7020.96) | 36010.7 (7362.59)
  C2D1: Endoglin (n= 3, 2, 6, 3, 4, 5, 5, 2, 20) | 22204.3 (1736.96) | 32984.2 (691.27) | 23247.5 (5843.99) | 27246.9 (4925.02) | 28478.7 (5527.04) | 24736.3 (5716.80) | 27295.5 (8538.87) | 27813.5 (15243.7) | 37263.6 (9744.94)
  C3D1: Endoglin (n= 3, 2, 4, 3, 1, 4, 3, 1, 12) | 24503.9 (3500.18) | 29688.2 (2138.72) | 24944.4 (2436.94) | 31266.8 (3466.76) | 22233.2 (NA) — Standard deviation was not reported since only 1 participant was evaluable for this arm group. | 24395.8 (2414.67) | 24540.0 (4547.98) | 33259.2 (NA) — Standard deviation was not reported since only 1 participant was evaluable for this arm group. | 35347.9 (6702.15)
  EOT: Endoglin (n= 5, 5, 2, 3, 4, 4, 5, 5, 17) | 28268.0 (7727.06) | 26852.1 (6037.41) | 23453.9 (3631.56) | 28064.5 (4097.50) | 28094.3 (1554.41) | 29350.8 (2213.84) | 38234.3 (16532.0) | 26855.9 (4711.30) | 35726.0 (8159.01)

22. Other Pre Specified Outcome: Soluble Protein Biomarker [Placental Growth Factor (PLGF), Transforming Growth Beta 1 (TGFB1), Vascular Endothelial Growth Factor A (VEGF-A)]: Part 1 and Part 2
Description: Plasma concentrations of soluble proteins (PLGF, TGFB1, VEGF-A) may be associated with tumor angiogenesis or tumor physiology and may correlate with efficacy or biological activity.
Time Frame: Baseline (pre-dose of C1D1), C1D1 6 hours post dosing, C1D22, C2D1, C3D1 and end of treatment (Day 490)
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | PF-03446962 0.5 mg/kg: Part 1 | PF-03446962 1 mg/kg: Part 1 | PF-03446962 2 mg/kg : Part 1 | PF-03446962 3 mg/kg: Part 1 | PF-03446962 4.5 mg/kg: Part 1 | PF-03446962 6.75 mg/kg: Part 1 | PF-03446962 10 mg/kg: Part 1 | PF-03446962 15 mg/kg: Part 1 | PF-03446962 7 mg/kg: Part 2
Number analyzed (Participants) | 5 | 5 | 6 | 3 | 4 | 8 | 6 | 5 | 24
pg/ml
  Baseline: PLGF (n=4, 3, 5, 3, 2, 7, 6, 5, 21) | 9.1 (5.69) | 9.3 (2.06) | 14.7 (4.30) | 6.4 (2.50) | 10.6 (1.98) | 13.4 (5.86) | 17.2 (9.83) | 22.3 (19.56) | 13.4 (5.27)
  C1D16H: PLGF (n=4, 3, 5, 3, 2, 7, 6, 5, 22) | 8.4 (1.56) | 6.1 (3.09) | 12.4 (2.94) | 6.4 (3.04) | 8.4 (1.91) | 8.7 (2.84) | 22.0 (25.07) | 15.0 (11.95) | 8.9 (3.66)
  C1D22: PLGF (n=4, 5, 6, 2, 3, 6, 6, 4, 18) | 11.3 (6.94) | 9.6 (3.98) | 9.5 (2.48) | 6.4 (0.85) | 6.6 (3.01) | 6.8 (2.19) | 13.6 (9.77) | 8.5 (1.89) | 8.4 (3.28)
  C2D1: PLGF (n=3, 2, 6, 1, 3, 4, 3, 2, 18) | 9.4 (4.81) | 7.6 (0.49) | 9.8 (3.55) | 11.0 (NA) — Standard deviation was not reported since only 1 participant was evaluable for this arm group. | 7.3 (3.00) | 9.7 (5.09) | 16.5 (13.95) | 7.1 (1.91) | 8.3 (2.39)
  C3D1: PLGF (n=3, 2, 3, 1, 1, 4, 2, 1, 10) | 11.0 (3.87) | 15.2 (5.66) | 9.9 (4.37) | 7.5 (NA) — Standard deviation was not reported since only 1 participant was evaluable for this arm group. | 11.9 (NA) — Standard deviation was not reported since only 1 participant was evaluable for this arm group. | 7.1 (2.05) | 8.9 (3.54) | 7.0 (NA) — Standard deviation was not reported since only 1 participant was evaluable for this arm group. | 6.9 (1.92)
  EOT: PLGF (n=5, 4, 2, 2, 2, 3, 2, 4, 14) | 11.8 (3.15) | 8.3 (3.20) | 8.7 (0.64) | 8.6 (1.34) | 6.8 (3.39) | 9.1 (2.29) | 20.1 (12.45) | 19.9 (20.49) | 7.8 (3.30)
  Baseline: TGFb1 (n=5, 5, 6, 3, 4, 8, 7, 6, 24) | 192856 (167465) | 58530.3 (70338.7) | 188182 (199702) | 322573 (249585) | 174960 (171958) | 236277 (108993) | 190445 (113478) | 184332 (59292.8) | 72635.0 (69063.0)
  C1D16H: TGFb1 (n=4, 3, 6, 3, 4, 8, 7, 6, 24) | 185701 (107677) | 203200 (158543) | 225230 (129870) | 269437 (225974) | 297119 (87426.7) | 265679 (89033.4) | 311792 (104827) | 282944 (196959) | 66293.0 (47427.2)
  C1D22: TGFb1 (n=4, 5, 6, 3, 4, 6, 7, 5, 20) | 160128 (119814) | 328947 (271795) | 272123 (162239) | 307758 (206598) | 298611 (178683) | 234304 (146086) | 212425 (106195) | 340151 (232305) | 65483.2 (35965.8)
  C2D1: TGFb1 (n=3, 2, 6, 3, 4, 5, 5, 2, 20) | 216478 (33849.2) | 162468 (63111.4) | 182580 (112201) | 213943 (64818.6) | 302708 (213685) | 258286 (88746.3) | 230125 (174311) | 156793 (108469) | 65275.6 (48954.3)
  C3D1: TGFb1 (n=3, 2, 4, 3, 1, 4, 3, 1, 12) | 387504 (211630) | 327375 (208226) | 281413 (181027) | 191820 (123461) | 238304 (NA) — Standard deviation was not reported since only 1 participant was evaluable for this arm group. | 326939 (184808) | 295378 (133164) | 62172.4 (NA) — Standard deviation was not reported since only 1 participant was evaluable for this arm group. | 73118.3 (49778.0)
  EOT: TGFb1 (n=5, 5, 2, 3, 4, 4, 5, 5, 17) | 172056 (100831) | 279062 (214205) | 203631 (254400) | 292165 (163750) | 250882 (165972) | 336973 (225077) | 183926 (163333) | 486629 (381351) | 95074.9 (92796.5)
  Baseline: VEGF-A (n=4, 5, 6, 3, 3, 8, 7, 6, 24) | 907.5 (479.21) | 222.3 (201.48) | 452.5 (328.65) | 522.2 (512.23) | 669.4 (608.96) | 437.7 (268.81) | 538.9 (421.35) | 634.6 (874.12) | 613.5 (984.96)
  C1D16H: VEGF-A (n=4, 3, 6, 3, 4, 8, 7, 6, 24) | 988.3 (646.26) | 476.4 (155.58) | 788.6 (578.29) | 592.6 (684.51) | 587.5 (437.86) | 542.3 (400.82) | 648.7 (482.00) | 671.6 (997.74) | 671.1 (998.34)
  C1D22: VEGF-A (n=4, 5, 6, 3, 4, 6, 7, 4, 20) | 564.3 (212.89) | 772.5 (466.51) | 786.5 (650.76) | 748.0 (527.71) | 479.2 (359.29) | 617.6 (481.63) | 656.6 (579.52) | 1432.7 (1566.42) | 1078.9 (1095.02)
  C2D1: VEGF-A (n=3, 2, 6, 3, 4, 5, 5, 2, 20) | 623.7 (330.44) | 321.7 (401.42) | 608.8 (789.07) | 671.0 (349.68) | 600.0 (529.40) | 653.6 (339.01) | 754.8 (683.82) | 1904.2 (2559.16) | 1064.3 (2200.07)
  C3D1: VEGF-A (n=3, 2, 4, 3, 1, 4, 3, 1, 12) | 1106.9 (374.74) | 378.6 (427.52) | 633.0 (332.78) | 526.5 (324.46) | 710.1 (NA) — Standard deviation was not reported since only 1 participant was evaluable for this arm group. | 621.1 (409.65) | 980.7 (656.43) | 76.4 (NA) — Standard deviation was not reported since only 1 participant was evaluable for this arm group. | 641.8 (651.66)
  EOT: VEGF-A (n=5, 5, 2, 3, 4, 4, 5, 5, 17) | 991.3 (606.54) | 700.2 (406.16) | 231.6 (187.74) | 579.8 (205.68) | 511.0 (496.32) | 804.5 (577.55) | 1195.4 (1390.00) | 871.9 (1068.86) | 802.5 (880.22)

23. Other Pre Specified Outcome: Soluble Protein Biomarker [Vascular Endothelial Growth Factor C (VEGF-C), Vascular Endothelial Growth Factor-d (VEGF-d), Vascular Endothelial Growth Factor Receptor Type 1 (VEGFR1)]: Part 1 and Part 2
Description: Plasma concentrations of soluble proteins (VEGF-C, VEGF-d, VEGFR1) may be associated with tumor angiogenesis or tumor physiology and may correlate with efficacy or biological activity.
Time Frame: Baseline (pre-dose of C1D1), C1D1 6 hours post dosing, C1D22, C2D1, C3D1 and end of treatment (Day 490)
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | PF-03446962 0.5 mg/kg: Part 1 | PF-03446962 1 mg/kg: Part 1 | PF-03446962 2 mg/kg : Part 1 | PF-03446962 3 mg/kg: Part 1 | PF-03446962 4.5 mg/kg: Part 1 | PF-03446962 6.75 mg/kg: Part 1 | PF-03446962 10 mg/kg: Part 1 | PF-03446962 15 mg/kg: Part 1 | PF-03446962 7 mg/kg: Part 2
Number analyzed (Participants) | 5 | 5 | 6 | 3 | 4 | 8 | 7 | 6 | 24
pg/ml
  Baseline: VEGF-C (n= 3, 1, 3, 2, 2, 4, 4, 4, 15) | 157.8 (47.72) | 129.4 (NA) — Standard deviation was not reported since only 1 participant was evaluable for this arm group. | 80.8 (26.11) | 130.1 (74.10) | 200.7 (55.58) | 86.1 (25.17) | 85.5 (23.49) | 195.3 (164.87) | 123.1 (59.79)
  C1D16H: VEGF-C (n= 2, 2, 4, 2, 2, 5, 5, 4, 13) | 128.2 (82.17) | 41.8 (7.71) | 102.2 (27.40) | 146.0 (129.90) | 151.4 (67.03) | 116.9 (62.28) | 80.4 (24.55) | 120.2 (63.80) | 144.2 (40.73)
  C1D22: VEGF-C (n= 3, 5, 4, 2, 2, 4, 4, 4, 12) | 86.7 (58.88) | 85.7 (40.52) | 129.1 (129.05) | 82.3 (45.18) | 187.6 (8.84) | 103.8 (45.97) | 130.9 (78.92) | 193.8 (42.02) | 154.1 (85.63)
  C2D1: VEGF-C (n= 2, 1, 2, 1, 2, 4, 4, 1, 11) | 82.0 (56.92) | 102.8 (NA) — Standard deviation was not reported since only 1 participant was evaluable for this arm group. | 73.0 (27.37) | 75.5 (NA) — Standard deviation was not reported since only 1 participant was evaluable for this arm group. | 195.5 (22.56) | 78.1 (24.17) | 92.7 (60.15) | 209.0 (NA) — Standard deviation was not reported since only 1 participant was evaluable for this arm group. | 201.4 (91.96)
  C3D1: VEGF-C (n= 2, 1, 2, 0, 1, 3, 1, 0, 8) | 217.8 (175.08) | 139.8 (NA) — Standard deviation was not reported since only 1 participant was evaluable for this arm group. | 100.2 (64.49) | NA (NA) — Data was not reported since no participant was evaluable for this arm group | 72.5 (NA) — Standard deviation was not reported since only 1 participant was evaluable for this arm group. | 93.6 (38.86) | 90.5 (NA) — Standard deviation was not reported since only 1 participant was evaluable for this arm group. | NA (NA) — Data was not reported since no participant was evaluable for this arm group | 190.5 (71.75)
  EOT: VEGF-C (n= 5, 4, 0, 1, 2, 3, 4, 5, 10) | 140.0 (102.64) | 110.1 (55.86) | NA (NA) — Data was not reported since no participant was evaluable for this arm group | 60.1 (NA) — Standard deviation was not reported since only 1 participant was evaluable for this arm group. | 146.8 (108.75) | 131.8 (21.49) | 138.0 (112.15) | 114.9 (43.61) | 186.1 (91.79)
  Baseline: VEGF-d (n= 5, 5, 6, 3, 4, 8, 7, 6, 24) | 1482.0 (661.38) | 2365.6 (2277.70) | 1694.0 (1200.02) | 1393.9 (371.40) | 2073.3 (1258.05) | 2421.0 (2415.95) | 1282.9 (308.22) | 1144.6 (214.88) | 2127.8 (1620.79)
  C1D16H: VEGF-d (n= 4, 3, 6, 3, 4, 8, 7, 6, 24) | 1521.1 (863.10) | 1554.8 (968.88) | 1862.7 (1422.39) | 1453.6 (469.17) | 1400.7 (634.61) | 2638.6 (3254.13) | 1487.3 (654.83) | 1031.1 (285.11) | 2142.8 (1494.28)
  C1D22: VEGF-d (n= 4, 5, 6, 3, 4, 6, 7, 5, 19) | 896.2 (257.64) | 1544.2 (952.69) | 1627.6 (1133.17) | 1376.2 (468.11) | 1916.3 (1499.55) | 2831.2 (3980.28) | 1634.0 (741.59) | 1191.6 (407.20) | 2375.2 (1506.25)
  C2D1: VEGF-d (n= 3, 2, 6, 3, 4, 5, 5, 2, 20) | 1276.2 (830.02) | 1787.2 (1467.67) | 1873.7 (1363.68) | 1359.8 (590.91) | 2277.6 (2283.70) | 2557.3 (3427.60) | 1333.5 (404.55) | 1025.5 (132.44) | 1957.2 (963.83)
  C3D1: VEGF-d (n= 3, 2, 4, 3, 1, 4, 3, 1, 12) | 1259.9 (763.65) | 1826.2 (1660.36) | 1954.2 (1737.30) | 1300.9 (623.64) | 1584.0 (NA) — Standard deviation was not reported since only 1 participant was evaluable for this arm group. | 3876.5 (5419.26) | 1100.3 (395.55) | 1470.1 (NA) — Standard deviation was not reported since only 1 participant was evaluable for this arm group. | 2094.4 (837.78)
  EOT: VEGF-d (n= 5, 5, 2, 3, 4, 4, 5, 5, 17) | 1259.0 (640.63) | 1463.6 (813.87) | 2218.0 (2141.83) | 1289.9 (633.94) | 2181.2 (1622.16) | 2079.0 (1987.67) | 1464.0 (959.39) | 1093.7 (308.36) | 2011.1 (988.62)
  Baseline: VEGFR1 (n= 5, 5, 6, 3, 4, 7, 7, 6, 23) | 1377.6 (2854.50) | 216.1 (302.01) | 118.1 (65.01) | 75.3 (20.82) | 262.3 (261.24) | 77.5 (39.81) | 219.5 (195.62) | 200.4 (119.61) | 243.6 (128.59)
  C1D16H: VEGFR1 (n= 4, 3, 6, 3, 4, 8, 6, 6, 23) | 98.6 (45.70) | 230.0 (262.82) | 200.2 (241.23) | 258.4 (336.53) | 656.3 (1160.02) | 79.6 (62.56) | 362.6 (525.74) | 134.8 (83.44) | 251.7 (306.54)
  C1D22: VEGFR1 (n= 4, 5, 6, 3, 3, 5, 7, 4, 20) | 102.1 (40.47) | 325.0 (545.00) | 181.8 (207.89) | 79.2 (27.82) | 377.0 (372.66) | 77.8 (30.55) | 127.9 (91.93) | 149.3 (95.67) | 187.6 (80.10)
  C2D1: VEGFR1 (n= 3, 1, 6, 3, 4, 5, 5, 2, 20) | 63.0 (24.69) | 1556.8 (NA) — Standard deviation was not reported since only 1 participant was evaluable for this arm group. | 464.1 (611.85) | 81.9 (37.78) | 215.9 (236.35) | 56.4 (22.50) | 179.1 (153.00) | 164.5 (89.31) | 656.5 (2066.54)
  C3D1: VEGFR1 (n= 3, 2, 4, 3, 1, 4, 2, 1, 12) | 97.7 (45.58) | 2659.5 (3611.41) | 109.5 (34.95) | 244.4 (304.26) | 386.2 (NA) — Standard deviation was not reported since only 1 participant was evaluable for this arm group. | 50.3 (26.44) | 388.4 (351.79) | 283.3 (NA) — Standard deviation was not reported since only 1 participant was evaluable for this arm group. | 236.1 (245.35)
  EOT: VEGFR1 (n= 5, 5, 2, 2, 4, 4, 4, 5, 17) | 125.2 (57.71) | 316.4 (561.02) | 412.9 (389.40) | 209.0 (148.00) | 173.1 (110.45) | 118.9 (22.12) | 365.3 (267.06) | 175.3 (138.87) | 242.4 (140.35)

24. Other Pre Specified Outcome: Soluble Protein Biomarker [Vascular Endothelial Growth Factor Receptor Type 2 (VEGFR2), Vascular Endothelial Growth Factor Receptor Type 3 (VEGFR3)]: Part 1 and Part 2
Description: Plasma concentrations of soluble proteins (VEGFR2, VEGFR3) may be associated with tumor angiogenesis or tumor physiology and may correlate with efficacy or biological activity.
Time Frame: Baseline (pre-dose of C1D1), C1D1 6 hours post dosing, C1D22, C2D1, C3D1 and end of treatment (Day 490)
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | PF-03446962 0.5 mg/kg: Part 1 | PF-03446962 1 mg/kg: Part 1 | PF-03446962 2 mg/kg : Part 1 | PF-03446962 3 mg/kg: Part 1 | PF-03446962 4.5 mg/kg: Part 1 | PF-03446962 6.75 mg/kg: Part 1 | PF-03446962 10 mg/kg: Part 1 | PF-03446962 15 mg/kg: Part 1 | PF-03446962 7 mg/kg: Part 2
Number analyzed (Participants) | 5 | 5 | 6 | 3 | 4 | 8 | 7 | 6 | 24
pg/ml
  Baseline: VEGFR2 (n= 5, 5, 6, 3, 4, 8, 7, 6, 24) | 8414.2 (3145.86) | 8281.8 (4500.81) | 8834.8 (1749.43) | 10475.6 (862.91) | 9536.4 (2527.39) | 7526.1 (1910.18) | 7712.5 (2738.41) | 8934.9 (1266.00) | 6495.9 (2172.45)
  C1D16H: VEGFR2 (n= 4, 3, 6, 3, 4, 8, 7, 6, 24) | 7989.8 (3208.34) | 7069.9 (5395.12) | 9884.4 (3258.50) | 10980.4 (1881.48) | 7707.1 (2003.97) | 7902.7 (2606.45) | 7500.6 (2409.88) | 8827.1 (1458.20) | 6708.1 (2314.78)
  C1D22: VEGFR2 (n= 4, 5, 6, 3, 4, 6, 7, 5, 20) | 8310.6 (4171.13) | 9672.8 (4841.31) | 9057.3 (1614.38) | 10248.0 (1886.86) | 8057.2 (1948.44) | 8912.0 (2327.17) | 9230.3 (4272.69) | 9572.0 (2736.01) | 7147.6 (2735.63)
  C2D1: VEGFR2 (n= 3, 2, 6, 3, 4, 5, 5, 2, 20) | 6699.4 (3398.50) | 9896.8 (1626.91) | 9191.5 (2061.89) | 9354.7 (2102.62) | 6621.2 (1637.27) | 8016.8 (1689.68) | 7727.3 (3137.81) | 8567.2 (222.95) | 7468.4 (2757.65)
  C3D1: VEGFR2 (n= 3, 2, 4, 3, 1, 4, 3, 1, 12) | 8780.4 (4855.85) | 9372.8 (1111.71) | 9736.1 (1396.40) | 9988.4 (1704.87) | 7180.0 (NA) — Standard deviation was not reported since only 1 participant was evaluable for this arm group. | 9289.2 (2003.70) | 9784.5 (2193.47) | 9632.8 (NA) — Standard deviation was not reported since only 1 participant was evaluable for this arm group. | 7087.9 (2430.45)
  EOT: VEGFR2 (n= 5, 5, 2, 3, 4, 4, 5, 5, 17) | 9541.6 (3903.58) | 8297.5 (4291.01) | 7490.4 (5124.26) | 11521.7 (1822.45) | 8151.8 (2508.61) | 10018.0 (2860.16) | 7771.7 (3593.10) | 9357.8 (2845.47) | 8151.0 (2254.12)
  Baseline: VEGFR3 (n= 5, 5, 6, 3, 4, 8, 7, 6, 24) | 421297 (89735.8) | 396991 (111696) | 340605 (106111) | 282449 (52144.0) | 336510 (183465) | 402326 (127490) | 377133 (109330) | 409280 (166548) | 423268 (152555)
  C1D16H: VEGFR3 (n= 4, 3, 6, 3, 4, 8, 7, 6, 24) | 403555 (118261) | 417915 (101370) | 376867 (146099) | 282590 (58032.4) | 301990 (114920) | 371861 (130334) | 361958 (106007) | 375385 (89006.0) | 427567 (133307)
  C1D22: VEGFR3 (n= 4, 5, 6, 3, 4, 6, 7, 5, 20) | 418199 (135460) | 413223 (111775) | 482016 (227736) | 278094 (29688.1) | 335397 (159853) | 405426 (135402) | 384832 (157842) | 367493 (104354) | 439596 (117856)
  C2D1: VEGFR3 (n= 3, 2, 6, 3, 4, 5, 5, 2, 20) | 456367 (205119) | 283799 (30962.7) | 483165 (166891) | 299955 (42094.9) | 326823 (171815) | 403432 (164005) | 326291 (81142.0) | 330917 (3323.61) | 436507 (130015)
  C3D1: VEGFR3 (n= 3, 2, 4, 3, 1, 4, 3, 1, 12) | 486756 (156161) | 335446 (688.51) | 380689 (189516) | 272982 (12015.1) | 563837 (NA) — Standard deviation was not reported since only 1 participant was evaluable for this arm group. | 356012 (127436) | 301489 (85606.4) | 309162 (NA) — Standard deviation was not reported since only 1 participant was evaluable for this arm group. | 401286 (120518)
  EOT: VEGFR3 (n= 5, 5, 2, 3, 4, 4, 5, 5, 17) | 456664 (83808.5) | 358829 (70878.1) | 396443 (324477) | 306684 (72478.1) | 319223 (117705) | 419244 (54326.1) | 446291 (293311) | 440490 (118906) | 457457 (144474)

25. Other Pre Specified Outcome: Circulating Endothelial Cells (CEC)and Circulating Endothelial Progenitors (CEP): Part 1 and Part 2
Description: Circulating endothelial cells (CECs) are noninvasive marker of vascular damage, remodeling, and dysfunction. Blood samples for the assessment of CECs and circulating CEPs were collected to analyze effects of therapy on the number, viability/apoptotic state, and/or target activity/expression in CECs. Circulating Cells were classified as CEPs if cluster differentiation 133 positive cells (CD133+) were detected.
Time Frame: Baseline (pre-dose of C1D1), C1D1 6 hours post dosing, C1D22, C2D1, C3D1 and end of treatment (Day 490)
Population: Data was reported in individual participant listings but not statistically summarized due to statistical constraints.
Arm/Group | PF-03446962 0.5 mg/kg: Part 1 | PF-03446962 1 mg/kg: Part 1 | PF-03446962 2 mg/kg : Part 1 | PF-03446962 3 mg/kg: Part 1 | PF-03446962 4.5 mg/kg: Part 1 | PF-03446962 6.75 mg/kg: Part 1 | PF-03446962 10 mg/kg: Part 1 | PF-03446962 15 mg/kg: Part 1 | PF-03446962 7 mg/kg: Part 2
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | PF-03446962
Serious Adverse Events (participants affected / at risk) | 24/68
Other Adverse Events (participants affected / at risk) | 68/68
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PF-03446962 (N=68)
Anaemia (Blood and lymphatic system disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 4
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Haematemesis (Gastrointestinal disorders) | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Condition aggravated (General disorders) | 1
Disease progression (General disorders) | 3
Fatigue (General disorders) | 1
Pyrexia (General disorders) | 2
Hepatitis acute (Hepatobiliary disorders) | 1
Hypersensitivity (Immune system disorders) | 1
Infection (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Blood albumin decreased (Investigations) | 1
Failure to thrive (Metabolism and nutrition disorders) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Tumour necrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Somnolence (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Suicide attempt (Psychiatric disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1
Embolism (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PF-03446962 (N=68)
Anaemia (Blood and lymphatic system disorders) | 5
Leukocytosis (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 10
Vertigo (Ear and labyrinth disorders) | 1
Conjunctival haemorrhage (Eye disorders) | 1
Eye discharge (Eye disorders) | 1
Eye pain (Eye disorders) | 1
Eyelid oedema (Eye disorders) | 2
Abdominal distension (Gastrointestinal disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 5
Abdominal pain lower (Gastrointestinal disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 6
Ascites (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 8
Diarrhoea (Gastrointestinal disorders) | 6
Melaena (Gastrointestinal disorders) | 1
Mouth haemorrhage (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 18
Rectal haemorrhage (Gastrointestinal disorders) | 1
Subileus (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 9
Asthenia (General disorders) | 17
Chills (General disorders) | 7
Fatigue (General disorders) | 19
Mucosal inflammation (General disorders) | 3
Oedema peripheral (General disorders) | 12
Pelvic mass (General disorders) | 1
Pyrexia (General disorders) | 12
Gallbladder disorder (Hepatobiliary disorders) | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 3
Hypertransaminasaemia (Hepatobiliary disorders) | 1
Portal vein thrombosis (Hepatobiliary disorders) | 1
Herpes simplex (Infections and infestations) | 1
Influenza (Infections and infestations) | 2
Rhinovirus infection (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 4
Skin infection (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 6
Urinary tract infection (Infections and infestations) | 3
Periorbital haematoma (Injury, poisoning and procedural complications) | 1
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 1
Ammonia increased (Investigations) | 1
Amylase increased (Investigations) | 8
Aspartate aminotransferase increased (Investigations) | 5
Blood alkaline phosphatase increased (Investigations) | 10
Blood bilirubin increased (Investigations) | 1
Blood creatinine increased (Investigations) | 5
Blood potassium increased (Investigations) | 1
Breath sounds abnormal (Investigations) | 1
Electrocardiogram QT prolonged (Investigations) | 3
Heart rate increased (Investigations) | 1
Laboratory test abnormal (Investigations) | 1
Lipase increased (Investigations) | 8
Liver function test abnormal (Investigations) | 1
Platelet count decreased (Investigations) | 8
Transaminases increased (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 12
Dehydration (Metabolism and nutrition disorders) | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 7
Hyperuricaemia (Metabolism and nutrition disorders) | 5
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2
Hypokalaemia (Metabolism and nutrition disorders) | 5
Hypomagnesaemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 5
Flank pain (Musculoskeletal and connective tissue disorders) | 2
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Ataxia (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 7
Dysgeusia (Nervous system disorders) | 1
Headache (Nervous system disorders) | 8
Paraesthesia (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 2
Confusional state (Psychiatric disorders) | 2
Sleep disorder (Psychiatric disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Proteinuria (Renal and urinary disorders) | 5
Renal failure acute (Renal and urinary disorders) | 1
Urinary incontinence (Renal and urinary disorders) | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1
Scrotal oedema (Reproductive system and breast disorders) | 1
Testicular oedema (Reproductive system and breast disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 14
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 2
Ecchymosis (Skin and subcutaneous tissue disorders) | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 4
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 4
Rash (Skin and subcutaneous tissue disorders) | 3
Skin lesion (Skin and subcutaneous tissue disorders) | 2
Swelling face (Skin and subcutaneous tissue disorders) | 1
Telangiectasia (Skin and subcutaneous tissue disorders) | 6
Hypertension (Vascular disorders) | 2
Hypotension (Vascular disorders) | 5
Intra-abdominal haematoma (Vascular disorders) | 1
Vasodilatation (Vascular disorders) | 1
Lymphopenia (Blood and lymphatic system disorders) | 1
Conjunctivitis (Eye disorders) | 2
Photopsia (Eye disorders) | 1
Vision blurred (Eye disorders) | 2
Vitreous floaters (Eye disorders) | 1
Dry mouth (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 2
Gastric haemorrhage (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Intestinal obstruction (Gastrointestinal disorders) | 1
Influenza like illness (General disorders) | 1
Pain (General disorders) | 1
Cytokine release syndrome (Immune system disorders) | 1
Multiple allergies (Immune system disorders) | 1
Cystitis (Infections and infestations) | 1
Fungal oesophagitis (Infections and infestations) | 1
Infection (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 2
Contusion (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 4
Aspartate aminotransferase (Investigations) | 1
Blood albumin decreased (Investigations) | 1
Blood calcium decreased (Investigations) | 1
Blood glucose increased (Investigations) | 1
Blood potassium decreased (Investigations) | 1
Blood pressure increased (Investigations) | 1
Blood sodium decreased (Investigations) | 1
Blood uric acid increased (Investigations) | 1
Creatinine renal clearance decreased (Investigations) | 1
Haemoglobin decreased (Investigations) | 4
Weight decreased (Investigations) | 1
Weight increased (Investigations) | 2
Hypernatraemia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 4
Groin pain (Musculoskeletal and connective tissue disorders) | 1
Muscle twitching (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Encephalopathy (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 1
Depression (Psychiatric disorders) | 1
Psychotic disorder (Psychiatric disorders) | 1
Dysuria (Renal and urinary disorders) | 1
Renal pain (Renal and urinary disorders) | 1
Pelvic pain (Reproductive system and breast disorders) | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1
Erythema (Skin and subcutaneous tissue disorders) | 2
Night sweats (Skin and subcutaneous tissue disorders) | 1
Rash papular (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1
Jugular vein thrombosis (Vascular disorders) | 1

LIMITATIONS AND CAVEATS:
Results for tumor vascular function adopting dynamic contrast enhanced-magnetic resonance imaging (DCE-MRI) was not reported as per change in planned analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.